CLINICAL TRIAL: NCT03214562
Title: A Phase 1b/2 Study of the BCL-2 Inhibitor Venetoclax in Combination With Standard Intensive AML Induction/Consolidation Therapy With FLAG-IDA in Patients With Newly Diagnosed or Relapsed/Refractory AML
Brief Title: Venetoclax With Combination Chemotherapy in Treating Patients With Newly Diagnosed or Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0979; NCI-2018-01119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0979 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: High Risk Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Idarubicin; pegfilgrastim; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, FLAG-IDA) (Experimental): See detailed description.
  Interventions: Drug: Cytarabine; Biological: Filgrastim; Drug: Fludarabine; Drug: Idarubicin; Biological: Pegfilgrastim; Drug: Venetoclax

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trial studies the best dose and side effects of venetoclax and how well it works when given with combination chemotherapy in treating patients with newly diagnosed acute myeloid leukemia or acute myeloid leukemia that has come back or does not respond to treatment. Venetoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine, cytarabine, filgrastim and idarubicin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax together with combination chemotherapy may work better in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability and to determine the dose-limiting toxicity and the maximum tolerated dose MTD of the combination of fludarabine, cytarabine, filgrastim (GCSF), idarubicin (FLAG-IDA) + venetoclax for patients with acute myeloid leukemia (AML) (Phase 1b).

II. To determine the overall activity of this combination in patients newly diagnosed or relapsed/refractory (AML) (Phase 2).

SECONDARY OBJECTIVES:

I. Determine the preliminary assessment of efficacy by response to revised International Working Group (IWG) criteria and time to response variables including overall survival (OS), event-free survival (EFS) and duration of response (DOR).

II. Determine biomarkers that may be predictive of venetoclax activity.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

INDUCTION THERAPY: Patients receive venetoclax orally (PO) on days 1-14, fludarabine intravenously (IV) over 30 minutes on days 2-6, cytarabine IV over 4 hours on days 2-6, idarubicin IV over 15-30 minutes on days 4 and 5, filgrastim subcutaneously (SC) on days 1-7, or pegfilgrastim SC after day 5. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients receive venetoclax PO on days 1-7, fludarabine IV over 30 minutes on days 2-4, cytarabine IV over 4 hours on days 2-4, filgrastim SC on days 1-7, or pegfilgrastim SC after days 3. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may also receive idarubicin as in Induction Therapy during 1 cycle of Consolidation Therapy per the treating physician.

MAINTENANCE THERAPY: Patients receive venetoclax PO on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML by World Health Organization (WHO) criteria. Patients with high risk myelodysplastic syndrome (MDS) as defined by the presence of >= 10% blasts are also eligible at the discretion of the principal investigator
* Patients older than 65 who are deemed fit to receive intensive chemotherapy by the treating physician will be eligible after discussion with the principal investigator (PI).
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Creatinine clearance >= 30 mL/min based on the Cockcroft-Gault equation
* Total bilirubin < 1.5 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement
* Ability to understand and provide signed informed consent
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug
* Only patients who are relapsed, refractory, or intolerant of standard AML therapy will be eligible for Part 1 (minimum of 1 prior line of AML-directed therapy)

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Patients having received any prior BCL2 inhibitor therapy
* Subject has known active central nervous system (CNS) involvement with AML
* Patients with New York Heart Association (NYHA) class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 40% by echocardiogram or multi-gated acquisition (MUGA) scan
* Patients with a history of myocardial infarction within the last 6 months or unstable / uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias
* Patients with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C
* Patients with known dysphagia, short-gut syndrome, or other conditions that would affect the ingestion or gastrointestinal absorption of drugs administered orally
* Subject has any other significant medical or psychiatric history that in the opinion of the investigator would adversely affect participation in this study
* Subject has a white blood cell count > 25 x 10{9}/L. (Note: hydroxyurea is permitted to meet this criterion)
* Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (a) appropriate method(s) of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double barrier methods (for example a condom in combination with a spermicide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 6 years
  Defined as complete response (CR) + CR with incomplete blood count recovery (CRi) + partial response (PR). Will be estimated along with the 95% credible interval.
CR/CRi rate | Up to 6 years
  Will be estimated along with the 95% credible interval.
Hematologic response | Up to 6 years
  Will be estimated along with the 95% credible interval.
Duration of response | From the date of initial response, assessed up to 6 years
  Defined as the number of days from the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first. Will be calculated for all patients.
Event-free survival | From the date of treatment initiation, assessed up to 6 years
  Defined as the number of days from the date of treatment initiation (i.e., course 1 day 1) to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first. Will be calculated for all patients. Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.
Overall survival | Up to 6 years
  Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.
Anti-tumor activity | Up to 6 years
  Will be summarized graphically and with descriptive statistics.
Pharmacodynamic markers | Up to 6 years
  Two samples t-test /Wilcoxon rank sum tests will be used to compare pharmacodynamics/pharmacokinetics (PD/PK) parameters between responder and non-responders, and logistic regression analysis will also be used to evaluate the association of PD/PK parameters with response.
Drug exposure levels | Up to 6 years
  Will be summarized graphically and with descriptive statistics.
Overall incidence and severity of all adverse events | Up to 6 years
  Graded using Common Toxicity Criteria version 4.0. Safety data will be summarized using frequency and percentage, by category and severity.

SECONDARY OUTCOMES:
Morphologic leukemia-free state | Up to 6 years
  Will be estimated along with the 95% credible interval.

OTHER OUTCOMES:
Exploratory biomarkers | Up to 6 years
  Will be summarized graphically and with descriptive statistics. Peripheral blood and bone marrow aspirate samples will be obtained at study specified time points. Biomarker assays may include, but are not limited to, BH3 profiling and characterization of BCL-2 and related proteins, and assessment of the depth of response and monitoring of disease recurrence by assessment of minimal residual disease (MRD) in the bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] DiNardo CD, Jen WY, Takahashi K, Kadia TM, Loghavi S, Daver NG, Xiao L, Reville PK, Issa GC, Short NJ, Sasaki K, Wang SA, Mullin JK, Pierce S, Bradley C, Borthakur G, Maiti A, Alvarado Y, Pemmaraju N, Ferrajoli A, Swaminathan M, Ohanian M, Abbas HA, Hammond D, Burger J, Haddad F, Montalban-Bravo G, Chien K, Masarova L, Yilmaz M, Jain N, Andreeff M, Garcia-Manero G, Kornblau S, Ravandi F, Jabbour E, Konopleva MY, Kantarjian HM. Long term results of venetoclax combined with FLAG-IDA induction and consolidation for newly diagnosed and relapsed or refractory acute myeloid leukemia. Leukemia. 2025 Apr;39(4):854-863. doi: 10.1038/s41375-025-02531-8. Epub 2025 Feb 25. PMID 40000842
- See also: M D Anderson Cancer Center — http://www.mdanderson.org